CLINICAL TRIAL: NCT06250517
Title: Impact of the Ex-vivo Pulmonary Perfusion System on the Microbiome of Lung Grafts and Their Inflammatory Reaction.
Acronym: ExBioma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vall d'Hebron Institute Research (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Irene Bello, Professor, Vall d'Hebron Institute Research
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ExBioma
Record Dates: First submitted 2023-12-23; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Lung Transplant Failure
MeSH Terms: interventions — Cryopreservation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVLP (Experimental)
  Interventions: Device: EVLP
- Cold preservation (Active Comparator)
  Interventions: Device: Cold preservation

INTERVENTIONS:
Device: EVLP — The right lung will be perfused for 3h with EVLP
  Arms: EVLP
Device: Cold preservation — The left lung will be cold preserved as usual protocol
  Arms: Cold preservation

SUMMARY:
It is known that the interactions of the graft and recipient microbiome are capable of modulating immune responses, inducing resilience or exacerbation of various inflammatory or fibrotic processes, therefore variations in the lung microbiome are associated with immunological changes in the transplanted lung.

The main objective is to understand the impact of new systems for conditioning and improving suboptimal lung grafts with ex vivo perfusion(EVLP) on the lung microbiome and its association with tissue inflammation.

The hypothesis is that manipulation of lung grafts and perfusion with broad-spectrum antibiotics during EVLP conditioning changes the lung microbiome, conditioning a less pro-inflammatory environment.

The methodology: This is a single-center prospective observational study. 7 consecutive brain-dead donors who do not meet the criteria to be lung donors will be included in the study. They will be carried out:

* P1. Detection: The donor without criteria to be a lung donor or rejected by all the transplant teams.
* P2. Extraction.
* P3. Cold preservation: The left lung will be cold-preserved
* P4. EVLP Conservation: The right lung will be prepared and conditioned for 3 hours using EVLP

The following samples will be taken at two times:

* T0: At the end of the extraction
* Bronchoalveolar lavage (BAL): Before tracheal clamping, BAL will be taken from the left main bronchus using bronchoscopy. The BAL will be performed on the right lung just before starting P4.
* Lung biopsy: Lung biopsy of the lower lobe of both grafts will be performed
* Preservation liquid or Perfusion liquid: 20 mL of preservation liquid that is in contact with the left graft before storage, as a sterility control (P3) and 20 mL of perfusion liquid before conditioning, as a sterility control (P4).
* T1: At the end of the conservation protocols (P3 or P4).
* B.A.L.
* Lung biopsy: left lower lobe.
* Preservation liquid or Infusion liquid: 20 mL of preservation liquid that is in contact with the left graft or 20 mL of perfusion fluid.

Due to the manipulation of the grafts during extraction and use of the technique, which involves extubating the donor and subsequently intubated again the grafts, as well as perfusion for a minimum of 3 hours with antibiotics, the use of EVLP could alter the microbiome of the grafts. This alteration could impact the obtaining of viable organs for transplant, in the immediate postoperative period as well as in the long-term results. There are no studies that analyse the change in the microbiome after conditioning with EVLP or its relationship with inflammatory parameters.

DETAILED DESCRIPTION:
SAMPLE TAKING AND STORAGE

* BAL:
* Technique: The bronchoscope will be inserted in segment 6, aliquots of sterile saline will be instilled. The procedure will be repeated in segments 3 and 5, in the case of the right lung, and in segment 6 and lingula in the left lung. 20-30cc of BAL will be completed for each graft.
* Storage: Samples will be frozen immediately after collection and transferred to the laboratory with a cold accumulator to ensure that they do not thaw.
* Analysis: The lung microbiome will be analysed.
* Lung biopsy:
* Technique: Lung biopsy of a minimum of 2cm3 will be taken using non-absorbable automatic suture.
* Storage: Samples will be preserved in RNA Stabilization solution Reagent (QIAGEN), which allows specimens to be kept at room temperature until frozen, avoiding RNA degradation.
* Analysis: RNA sequencing of transcription of inflammatory signals.
* Ex vivo perfusion liquid solution:
* Technique: Taking samples sterile with a 20cc syringe.
* Storage: Samples will be frozen immediately after collection and transferred to the laboratory with a cold accumulator to ensure that they do not thaw.
* Analysis: Microbiome analysis
* Preservation liquid solution:
* Technique: Taking samples sterile with a 20cc syringe.
* Storage: Samples will be frozen immediately after collection and transferred to the laboratory with a cold accumulator to ensure that they do not thaw.
* Analysis: Microbiome and cytokine analysis

All samples will be stored in a freezer at -80

- Microbiome analysis For the analysis of microbial diversity, the V4 variable region of the 16S gene will be amplified from bacterial DNA by PCR. Amplicons will be sequenced using Illumina (MiSeq) technology. Samples will be processed and more than 10,000 300bp sequences per sequence per sample will be generated.

Gene expression analysis RNA extraction will be performed using the commercial RNeasy Mini Kit (QIAGEN). Gene expression analysis will be performed by quantitative PCR (qPCR) using the predesigned TransplantRejection panel from SignArray (AnyGenes®, Paris, France) that includes 84 genes that have been described to be related to the immune response in transplant rejection. These are: Genes included in the panel: CX3CR1, ICAM1, ITGA2, ITGAE, ITGAM, PECAM1, THBS1, THBS2, VCAM1, COL1A2, CCR5, CCR7, CD40, CD40LG, CD80, CD86, CTLA4, CXCR3, STAT4, TGFB1, CD44 , CTGF, MMP1, MMP2, MMP7, MMP9, BMP7, CCL11, CCL2, CCL3, CCL4, CCL5, CSF2, CXCL10, IFNG, IL10, IL12A, IL13, IL16, IL1B, IL2, IL2RA, IL3, IL32, IL4, IL5 , IL6, IL8, TNF, TGFB2, TGFB3, TIMP1, VEGFA, MS4A1, CXCL11, CXCL9, CXCR4, ADAM17, C3, CASP1, CASP3, CASP8, CCR2, CCR3, CD14, CD28, CD8A, FAS, FASLG, FCGR1A, GZMA , GZMB, NFKB1, NOS2, PRF1, PSMB9, STAT1, STAT6, TAP1, TLR3, TLR4, TLR9, TNFAIP3, TNFSF10.

- Cytokine analysis The determination of cytokines in the perfusion fluid will be carried out using immunoassays based on Luminex™ xMAP™ technology (multi-analyte profiling) that allow the simultaneous quantification and detection of different secreted proteins (cytokines, chemokines, growth factors, etc.) We will use panels designed specifically for the gene products of interest.

Cytokine levels are measured using an immunoassay based on Luminex™ xMAP™ technology that allows for multi parametric analysis of the different cytokines. To this end, a personalized cytokine panel is designed based on the published literature on the effect of statins on the production of cytokines and other proinflammatory chemokines at a systemic level, as well as bibliographic evidence on the cytokines involved in lung transplantation. The cytokines analysed in the panel designed for this purpose are IFN gamma, IL-1 beta, IL-6, IL-8 (CXCL8), IL-18, IP-10 (CXCL10), MCP-1 (CCL2), MIP- 1 alpha (CCL3), TNF alpha, VEGF-D (Custom Procartaplex Multiplex Panel, Invitrogen, ThermoFisher Scientific, MA, USA). The immunological analysis will be carried out using the Invitrogen ProcartaPlex Analyst 1.0 software, supplied with the reagents.

- Bioinformatic analysis of the sequences To obtain the microbial composition of each sample, we will use the QIIME software. QIIME is a software pipeline that uses phylogenetic information and multivariate statistical techniques to compare microbial communities and determine, for example, whether they are statistically different. The program also identifies the species that contribute the most to these differences and discovers patterns of various types that characterize specific groups of samples.

ELIGIBILITY:
Inclusion Criteria:

* brain-death donors and donors after cardio circulatory death rejected for lung transplantation

Exclusion Criteria:

* Unilateral pneumonia
* Lack of consent for the donor's family.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in individual operational taxonomic units (OTUs) in lung parenchyma after the exvivo lung perfusion during 3 hours | After 3 hours of perfusion in ex vivo lung perfusion
  Analyse the lung microbiome and alpha diversity before the use of exvivo lung perfusion and after compared the micrological samples
Analysing with quantitative PCR of the genetic expression of 84 genes related to immune response in lung transplantation after the lung perfusion during 3h in exvivo lung perfusion system. | After 3 hours of perfusion in ex vivo lung perfusion
  Analyse with quantitative PCR of the genetic expression of 84 genes related with immune response in lung transplantation: CX3CR1, ICAM1, ITGA2, ITGAE, ITGAM, PECAM1, THBS1, THBS2, VCAM1, COL1A2, CCR5, CCR7, CD40, CD40LG, CD80, CD86, CTLA4, CXCR3, STAT4, TGFB1, CD44, CTGF, MMP1, MMP2, MMP7, MMP9, BMP7, CCL11, CCL2, CCL3, CCL4, CCL5, CSF2, CXCL10, IFNG, IL10, IL12A, IL13, IL16, IL1B, IL2, IL2RA, IL3, IL32, IL4, IL5, IL6, IL8, TNF, TGFB2, TGFB3, TIMP1, VEGFA, MS4A1, CXCL11, CXCL9, CXCR4, ADAM17, C3, CASP1, CASP3, CASP8, CCR2, CCR3, CD14, CD28, CD8A, FAS, FASLG, FCGR1A, GZMA, GZMB, NFKB1, NOS2, PRF1, PSMB9, STAT1, STAT6, TAP1, TLR3, TLR4, TLR9, TNFAIP3, TNFSF10 in lung samples before the use of exvivo lung perfusion and after, comparing them
Analyse the concentration of inflammatory cytokines after exvivo lung perfusion | After 3 hours of perfusion in ex vivo lung perfusion
  Analyse the concentration of inflammatory cytokines: IFN gamma,IL-1 beta,IL-6,IL-8 (CXCL8),IL-18,IP-10 (CXCL10),MCP-1 (CCL2),MIP-1 alpha (CCL3), TNF alpha,VEGF-D, with Luminex xMAP technique, in perfusion solution before and after the use of exvivo lung perfusion and comparing them
Change in individual operational taxonomic units (OTUs) in lung parenchyma after cold storage | After 3 hours of cold storage
  Analyse the lung microbiome and alpha diversity before and after the cold storage and compare the micrological samples.
Analysing the concentration of inflammatory citokines after cold storage | After 3 hours of cold storage
  Analyse the concentration of inflammatory cytokines: IFN gamma,IL-1 beta,IL-6,IL-8 (CXCL8),IL-18,IP-10 (CXCL10),MCP-1 (CCL2),MIP-1 alpha (CCL3), TNF alpha,VEGF-D, with Luminex xMAP technique, in perfusion solution before and after the cold storage and comparing them
Analysing with quantitative PCR of the genetic expression of 84 genes related to immune response in lung transplantation after cold storage | After 3 hours of cold storage
  Analyse with quantitative PCR of the genetic expression of 84 genes related with immune response in lung transplantation: CX3CR1, ICAM1, ITGA2, ITGAE, ITGAM, PECAM1, THBS1, THBS2, VCAM1, COL1A2, CCR5, CCR7, CD40, CD40LG, CD80, CD86, CTLA4, CXCR3, STAT4, TGFB1, CD44, CTGF, MMP1, MMP2, MMP7, MMP9, BMP7, CCL11, CCL2, CCL3, CCL4, CCL5, CSF2, CXCL10, IFNG, IL10, IL12A, IL13, IL16, IL1B, IL2, IL2RA, IL3, IL32, IL4, IL5, IL6, IL8, TNF, TGFB2, TGFB3, TIMP1, VEGFA, MS4A1, CXCL11, CXCL9, CXCR4, ADAM17, C3, CASP1, CASP3, CASP8, CCR2, CCR3, CD14, CD28, CD8A, FAS, FASLG, FCGR1A, GZMA, GZMB, NFKB1, NOS2, PRF1, PSMB9, STAT1, STAT6, TAP1, TLR3, TLR4, TLR9, TNFAIP3, TNFSF10 in lung samples before and after the cold storage, comparing them

CONTACTS AND LOCATIONS:
Overall Officials: Irene Bello Rodríguez, Professor, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No